CLINICAL TRIAL: NCT03651154
Title: PRICE 2: A Phase 3 Randomized Controlled Trial of Phlebotomy Resulting in Controlled Hypovolemia to Prevent Blood Loss in Major Hepatic Resections
Brief Title: Hypovolemic Phlebotomy to Reduce Blood Transfusions in Major Hepatic Resections
Acronym: PRICE2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 502
Record Dates: First submitted 2018-07-06; First posted 2018-08-29 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Liver Neoplasms; Hepatectomy; Blood Transfusion; Blood Loss, Surgical
MeSH Terms: conditions — Liver Neoplasms; Blood Loss, Surgical

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypovolemic Phlebotomy (Experimental): Hypovolemic Phlebotomy will consist of the withdrawal of 7-10 mL/kg of whole blood from the patient, as tolerated (e.g. for a 70kg patient, 490 to 700 mL of whole blood will be removed) The volume of removed blood will not be replaced by the administration of intravenous fluids.
  Removed blood will be transfused back to participant at the end of surgery. The phlebotomized whole blood will be transfused back after liver transection regardless of blood loss.
  Interventions: Procedure: Hypovolemic Phlebotomy
- Control (Standard of Care) (No Intervention): Standard of care (low CVP surgery). In this arm, standard anesthesia will be maintained.

INTERVENTIONS:
Procedure: Hypovolemic Phlebotomy — Removal of 7-10ml/kg of blood from participant, as tolerated after patient is under anesthesia, before liver resection start time
  Arms: Hypovolemic Phlebotomy

SUMMARY:
Major liver resection is associated with substantial intraoperative blood loss and subsequently blood transfusions. Blood transfusion in elective liver surgery is a significant factor of perioperative morbidity and mortality, as well as possibly long-term oncologic outcome. The purpose of this study is to use whole blood phlebotomy to decrease the central venous pressure, resulting in a state of relative hypovolemia. It is hypothesized that this intervention will lead to a decrease in blood loss at the time of liver resection and thus reduced blood transfusion in major liver surgeries.

DETAILED DESCRIPTION:
Major liver resection is associated with significant intraoperative blood loss and blood transfusions. Blood transfusion in elective liver surgery is a key determinant of perioperative morbidity and mortality, as well as possibly long-term oncologic outcome. Whole blood phlebotomy is a simple intervention, whose aim is to decrease the central venous pressure yielding a state of relative hypovolemia and thus lead to decreased blood loss and subsequently blood transfusion. Small studies, mostly from the liver transplant literature, would suggest that phlebotomy with controlled hypovolemia can result in decreased blood loss and blood transfusion. Since blood loss is an important issue in liver surgery, and the benefits of phlebotomy and controlled hypovolemia are unknown in liver resection patients, a rigorously conducted trial in a representative population of patients undergoing liver resection is warranted, and feasible. In this proposal, it is hypothesized that by the use of hypovolemic phlebotomy, it is possible to decrease blood loss and blood transfusions. To test this hypothesis the investigators plan to randomly allocate participants to hypovolemic phlebotomy plus standard of care or to standard of care. Participants will be those patients undergoing elective major liver resection at The Ottawa Hospital, le Centre Hospitalier de l'Université de Montréal, and le Centre Hospitalier de l'Université de Sherbrooke for any indication. The primary outcome will be red blood cells transfusion up to 30 days following surgery. Secondary outcomes will include intraoperative blood loss, other blood product transfusion requirements, perioperative morbidity and mortality, safety, physiologic parameters, and feasibility elements. A total of 440 patients will be randomized across the 3 sites in Ontario and Quebec. The efficacy of phlebotomy in terms of blood loss and transfusion prevention will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years)
* projected to undergo a major liver resection (≥3 segments resected or partially resected), a right posterior sectionectomy (segments 6/7), or central resection (4b/5) for any indication, or the resection of 1 or more segments in a known cirrhotic patient.

Exclusion Criteria:

* Age <18 years
* Preoperative hemoglobin <100g/L
* GFR clearance <60mL/min
* Abnormal coagulation parameters (not on warfarin and/or platelets count <100 X10^9/L)
* Evidence of hepatic metabolic disorder
* Active cardiac conditions: Unstable coronary syndromes; Severe valvular disease; and Myocardial infarction within 6 months prior to surgery
* History of significant cerebrovascular disease: Patients with clinically-significant stroke/CVA within the past 6 months or severe carotid stenosis (defined as >70%)
* History of significant peripheral vascular disease: Non-revascularized with regular/ongoing claudication
* Pregnancy
* Refusal of blood products
* Presence of active infection
* Preoperative autologous blood donation
* Planned intraoperative use of cell saver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2018-09-28 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Packed Red Blood Cell Transfusion Rates | 30 days post-operation
  Units of packed red blood cells transfused to participants

SECONDARY OUTCOMES:
Blood product transfusion rates | Postoperative setting up to 30 days following surgery
  Types and amount of other blood product transfusion rates in the 30 day period following surgery.
Intraoperative blood loss | up to 90 days before surgery; and on post-operative day 2
  Intraoperative blood loss is notoriously difficult to measure. It is suggested that calculation of blood loss using preoperative and postoperative hemoglobin levels in most consistently accurate. In order to minimize the risk of bias associated with any one method of intraoperative measurement of blood loss, three methods will be used independently. In the operating room, all blood and fluid aspirated from the abdomen will be measured accurately using graduated suction containers. As well, the amount of irrigation fluid will be carefully monitored and recorded. Finally, the weight of all surgical sponges will be measured. This information will be used by the surgeon and anesthesiologist to independently visually estimate blood loss, as is commonly done in clinical practice. In parallel, intraoperative blood loss will also be calculated based on an equation.
Perioperative morbidity and mortality | Postoperative setting up to 30 days following surgery
  Perioperative morbidity is assessed using the Dindo-Clavien scale and is defined as any deviation from the normal post-operative course. The scale (1-5) indicates the severity of an adverse event; where 1 is low (i.e. "any deviation from normal postoperative course without the need for intervention") and 5 means death of the patient (i.e. mortality).
Changes in physiologic parameters (Central Venous Pressure) | measured during surgery (intraoperatively)
  Central venous pressure (CVP) is a physiologic parameter that measures the blood pressure in the thoracic vena cava (in cm H20)
Changes in physiologic parameters (Pulse Pressure Variation) | measured during surgery (intraoperatively)
  Pulse Pressure variation (in %) is a predictor of fluid responsiveness

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Martel, MD, MSc, FRCSC, FACS, Principal Investigator — Ottawa Hospital Research Institute
Locations (4):
- Canada (4):
  - Vancouver General Hospital, Vancouver, British Columbia
  - The Ottawa Hospital, Ottawa, Ontario
  - Centre Hospitalier de l"Université de Sherbrooke, Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request, ethics approval and protocol approval from steering committee
Time Frame: Upon request during analysis
Access Criteria: Upon reasonable request, ethics approval and protocol approval from steering committee

REFERENCES:
- [Background] Sima CS, Jarnagin WR, Fong Y, Elkin E, Fischer M, Wuest D, D'Angelica M, DeMatteo RP, Blumgart LH, Gonen M. Predicting the risk of perioperative transfusion for patients undergoing elective hepatectomy. Ann Surg. 2009 Dec;250(6):914-21. doi: 10.1097/sla.0b013e3181b7fad3. PMID 19953711
- [Background] Alkozai EM, Lisman T, Porte RJ. Bleeding in liver surgery: prevention and treatment. Clin Liver Dis. 2009 Feb;13(1):145-154. doi: 10.1016/j.cld.2008.09.012. PMID 19150318
- [Background] Hallet J, Tsang M, Cheng ES, Habashi R, Kulyk I, Hanna SS, Coburn NG, Lin Y, Law CH, Karanicolas PJ. The Impact of Perioperative Red Blood Cell Transfusions on Long-Term Outcomes after Hepatectomy for Colorectal Liver Metastases. Ann Surg Oncol. 2015 Nov;22(12):4038-45. doi: 10.1245/s10434-015-4477-4. Epub 2015 Mar 10. PMID 25752895
- [Background] Bennett S, Baker LK, Martel G, Shorr R, Pawlik TM, Tinmouth A, McIsaac DI, Hebert PC, Karanicolas PJ, McIntyre L, Turgeon AF, Barkun J, Fergusson D. The impact of perioperative red blood cell transfusions in patients undergoing liver resection: a systematic review. HPB (Oxford). 2017 Apr;19(4):321-330. doi: 10.1016/j.hpb.2016.12.008. Epub 2017 Feb 1. PMID 28161216
- [Background] Massicotte L, Perrault MA, Denault AY, Klinck JR, Beaulieu D, Roy JD, Thibeault L, Roy A, McCormack M, Karakiewicz P. Effects of phlebotomy and phenylephrine infusion on portal venous pressure and systemic hemodynamics during liver transplantation. Transplantation. 2010 Apr 27;89(8):920-7. doi: 10.1097/TP.0b013e3181d7c40c. PMID 20216483
- [Background] Hashimoto T, Kokudo N, Orii R, Seyama Y, Sano K, Imamura H, Sugawara Y, Hasegawa K, Makuuchi M. Intraoperative blood salvage during liver resection: a randomized controlled trial. Ann Surg. 2007 May;245(5):686-91. doi: 10.1097/01.sla.0000255562.60215.3b. PMID 17457160
- [Background] Ryckx A, Christiaens C, Clarysse M, Vansteenkiste F, Steelant PJ, Sergeant G, Parmentier I, Pottel H, D'Hondt M. Central Venous Pressure Drop After Hypovolemic Phlebotomy is a Strong Independent Predictor of Intraoperative Blood Loss During Liver Resection. Ann Surg Oncol. 2017 May;24(5):1367-1375. doi: 10.1245/s10434-016-5737-7. Epub 2017 Jan 4. PMID 28054191
- [Background] Rekman J, Wherrett C, Bennett S, Gostimir M, Saeed S, Lemon K, Mimeault R, Balaa FK, Martel G. Safety and feasibility of phlebotomy with controlled hypovolemia to minimize blood loss in liver resections. Surgery. 2017 Mar;161(3):650-657. doi: 10.1016/j.surg.2016.08.026. Epub 2016 Oct 4. PMID 27712877
- [Derived] Martel G, Carrier FM, Wherrett C, Lenet T, Mallette K, Brousseau K, Monette L, Workneh A, Ruel M, Sabri E, Maddison H, Tokessy M, Wong PBY, Vandenbroucke-Menu F, Massicotte L, Chasse M, Collin Y, Perrault MA, Hamel-Perreault E, Park J, Lim S, Maltais V, Leung P, Gilbert RWD, Segedi M, Khalil JA, Bertens KA, Balaa FK, Ramsay T, Tinmouth A, Fergusson DA. Hypovolaemic phlebotomy in patients undergoing hepatic resection at higher risk of blood loss (PRICE-2): a randomised controlled trial. Lancet Gastroenterol Hepatol. 2025 Feb;10(2):114-124. doi: 10.1016/S2468-1253(24)00307-8. Epub 2024 Dec 9. PMID 39667380
- [Derived] Martel G, Lenet T, Wherrett C, Carrier FM, Monette L, Workneh A, Brousseau K, Ruel M, Chasse M, Collin Y, Vandenbroucke-Menu F, Hamel-Perreault E, Perreault MA, Park J, Lim S, Maltais V, Leung P, Gilbert RWD, Segedi M, Abou-Khalil J, Bertens KA, Balaa FK, Ramsay T, Fergusson DA. Phlebotomy resulting in controlled hypovolemia to prevent blood loss in major hepatic resections (PRICE-2): study protocol for a phase 3 randomized controlled trial. Trials. 2023 Jan 18;24(1):38. doi: 10.1186/s13063-022-07008-y. PMID 36653812